CLINICAL TRIAL: NCT00733317
Title: Phase 4 Study of Budesonide for Emergency Treatment of Acute Wheezing in Children
Brief Title: Budesonide for Emergency Treatment of Acute Wheezing in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kecioren Education and Training Hospital (Other)
Responsible Party: Principal Investigator, Cem Hasan Razi, MD, Kecioren Education and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B.10.0.İEG.0.11.00.01- 1864
Record Dates: First submitted 2008-08-12; First posted 2008-08-13 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-12

CONDITIONS: Asthma; Acute Asthma
Keywords: Wheezing; Acute asthma; Children; Budesonide; Emergency room
MeSH Terms: conditions — Asthma; Respiratory Sounds; Emergencies | interventions — Budesonide; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1-Budesonide nebulized suspension (Active Comparator): Children will receive 0.5 mg/ml budesonide nebules every 20 minutes for 3 times and will not give after 3 doses
  Interventions: Drug: 0.5 mg/ml budesonide nebules
- 2- 0.9% saline (Placebo Comparator): Children will receive 2 ml of saline every 20 minutes for 3 times and will not give after 3 doses
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: 0.5 mg/ml budesonide nebules — Children will receive 0.5 mg/ml budesonide nebules every 20 minutes for 3 times
  Other Names: Budesonide 0.5 mg/ml nebules
  Arms: 1-Budesonide nebulized suspension
Drug: Saline — Children will receive 2 ml of saline every 20 minutes for 3 times
  Other Names: 0.9% Saline solution
  Arms: 2- 0.9% saline

SUMMARY:
The purpose of this study is to determine if adding nebulized budesonide to the systemic steroid for treatment of acute wheezing has any additive benefit in the emergency room.

DETAILED DESCRIPTION:
Context: Inhaled steroids reduced admission rates in patients with acute asthma, but it is unclear if there is a benefit of inhaled corticosteroids when used in addition to systemic corticosteroids. There is insufficient evidence that inhaled corticosteroids result in clinically important changes in pulmonary function or clinical scores when used in acute asthma. Similarly, it was mentioned in the Cochrane Database of Systematic Reviews that further research is needed to clarify if there is a benefit of inhaled corticosteroids when used in addition to systemic steroids.

Objective: To determine if adding nebulized budesonide to the systemic steroid for treatment of acute wheezing in the emergency room has any benefit on, symptom score, hospitalization rate and time to discharge from emergency room.

Study Design/Setting/Participants: A double-blind, randomized, controlled trial of nebulized budesonide versus placebo for children 6 months to 6 years of age who have admitted to the emergency room for acute wheezing.

Intervention: Participants will receive standard therapy including SCS, albuterol, and ipratropium bromide and will be randomly assigned to also receive either nebulized BIS or saline.

Study Measures: Differences in asthma scores, vital signs, and the need for hospitalization will be compared between treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Children who have recurrent wheezing attacks and admitted to the emergency room for acute wheezing
* Pulmonary index score of 7-13
* Parental/guardian permission (informed consent) and if appropriate, child assent

Exclusion Criteria:

* Systemic corticosteroid use in the last 30 days
* Chronic lung diseases including cystic fibrosis
* Immunodeficiency
* Cardiac disease requiring surgery or medications
* Adverse drug reaction or allergy to budesonide, albuterol, ipratropium bromide, prednisone, prednisolone, or methylprednisolone
* Known renal or hepatic dysfunction
* Impending respiratory failure requiring positive pressure ventilation
* Immune deficiency
* Gastroesophageal reflux disease
* Suspected foreign body aspiration or croup
* Anatomic abnormalities of the respiratory tract

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2007-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Pulmonary index score at 2 to 4 hours | 2 to 4 hours

SECONDARY OUTCOMES:
Hospital admission rates | 4 hours
Proportion of subjects improving from severe to moderate, severe to mild, and moderate to mild. | 4 hours
Respiratory rate | 2 hours
Oxygen saturation | 2 hours
Time to discharge from the Emergency Department to home | 2 to 4 hours
Adverse reactions. | 2-5 days

CONTACTS AND LOCATIONS:
Overall Officials: C H Razi, MD, Study Director — Kecioren Education and Training Hospital; C H Razi, MD, Principal Investigator — Kecioren Education and Training Hospital
Locations (1):
- Kecioren Education and Training Hospital, Ankara, Kecioren, Turkey (Türkiye)